CLINICAL TRIAL: NCT06006273
Title: A Phase Ib Trial of Eribulin in Combination With Irinotecan and Temozolamide in Children With Relapsed or Refractory Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0163; NCI-2023-06570 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Refractory Solid Tumors
MeSH Terms: interventions — eribulin; Irinotecan; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A: Dose expansion-Ewings sarcoma (Experimental): The first group of participants in this phase will receive the highest dose of eribulin. Each group of participants enrolled after that will receive a slightly lower dose of the drug. Participants in this phase will be enrolled in 1 of 3 treatment arms, based on their disease type, and will receive the recommended dose combination found in the Dose Escalation phase.
  Interventions: Drug: Eribulin; Drug: Irinotecan; Drug: Temozolomide
- Arm B: Dose expansion -Rhabdomyosarcoma (Experimental): The first group of participants in this phase will receive the highest dose of eribulin. Each group of participants enrolled after that will receive a slightly lower dose of the drug. Participants in this phase will be enrolled in 1 of 3 treatment arms, based on their disease type, and will receive the recommended dose combination found in the Dose Escalation phase.
  Interventions: Drug: Eribulin; Drug: Irinotecan; Drug: Temozolomide
- Arm C: Dose expansion- other solid tumor histologies (Experimental): The first group of participants in this phase will receive the highest dose of eribulin. Each group of participants enrolled after that will receive a slightly lower dose of the drug. Participants in this phase will be enrolled in 1 of 3 treatment arms, based on their disease type, and will receive the recommended dose combination found in the Dose Escalation phase.
  Interventions: Drug: Eribulin; Drug: Irinotecan; Drug: Temozolomide
- Arm D: Dose finding levels 0,-1 and -2 (Experimental): The first group of participants in this phase will receive the highest dose of eribulin. Each group of participants enrolled after that will receive a slightly lower dose of the drug. Participants in this phase will be enrolled in 1 of 3 treatment arms, based on their disease type, and will receive the recommended dose combination found in the Dose Escalation phase.
  Interventions: Drug: Eribulin; Drug: Irinotecan; Drug: Temozolomide

INTERVENTIONS:
Drug: Eribulin — Given by vein (IV)
Drug: Irinotecan — Given by vein (IV)
Drug: Temozolomide — Given by PO

SUMMARY:
To find the recommended dose of eribulin that can be given in combination with irinotecan and temozolomide to treat relapsed and/or refractory solid tumors.

DETAILED DESCRIPTION:
Primary Objectives:

* To determine the maximum tolerated dose (MTD)/ recommended phase 2 dose (RP2D) of eribulin in combination with fixed doses of irinotecan and temozolomide.
* To determine the safety and tolerance of Eribulin when given in conjunction with Irinotecan and Temozolamide (IT) in children with refractory and relapsed (R/R) solid tumors.

Secondary Objectives:

--To observe and record disease response (anti-tumor activity). Although the clinical benefit of Eribulin when given together with Irinotecan and Temozolamide has not yet been established, the intent of offering this treatment is to provide a possible therapeutic benefit, and thus the patient will be carefully monitored for tumor response and symptom relief. Outcomes for disease response include Best Overall Response (BOR), Duration of Response (DOR), and Progression-Free Survival (PFS).

ELIGIBILITY:
Inclusion Criteria:

* Age: Patients must be > 1 year of age and ≤ 25 years of age at time of initiation of protocol therapy.
* Diagnosis: Patients have a histologically or radiographically confirmed relapsed or refractory solid tumor.
* Disease Status: Patients must have evaluable disease.
* Patients may have CNS metastases at study entry, if they are previously treated or stable (defined by not requiring initation or increased steroids for 7 days).
* Performance Level: Karnofsky ≥ 50% for patients >16 years old, and Lansky ≥ 50 for patients 1-16 years old. (Appendix I)
* Prior Therapy: Patients may have received prior therapy including single-agent irinotecan or temozolomide. Patients may not have previously been treated with combination therapy of irinotecan and temozolomide.
* Patients must be fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study.

  1. Hematopoietic growth factor: At least 7 days must have elapsed since the last administration of filgrastim, or 14 days since administration of pegfilgrastim.
  2. XRT: At least 7 days since the last dose of local palliative radiation therapy. Greater than 6 months must have elapsed since the last day of treatment if given total body irradiation, craniospinal irradiation.
  3. Autologous or Allogenic Stem Cell Transplant: Complete resolution of graft versus host disease and no current need for immunosuppressive medication. Greater than 3 months must have elapsed since engraftment and no longer requiring transfusion of platelets or injection of colony stimulating factors.

     * Organ Function Requirements
* Bone Marrow Function:

  1. Peripheral absolute neutrophil count (ANC) ≥ 750/µL
  2. Platelet count ≥ 75,000/µL (no platelet transfusion within 7 days prior to obtaining laboratory result)
* Adequate Renal Function:

  a. Creatinine clearance or glomerular filtration rate ≥ 70ml/min/1.73m2 (calculated or measured as appropriate for age and level of concern by treating MD)
* Adequate Liver Function:

  1. Total bilirubin ≤ 1.5x upper limit of normal (ULN) for age
  2. SGPT (ALT) ≤ 3 x ULN
  3. Serum albumin ≥ 2gm/dL Due to the risk of hepatic injury, including fatal hepatic failure, temozolomide should not be administered if total bilirubin is >2.0 mg/dl or SGPT(ALT)> 3 x ULN.

Informed Consent: All patients ≥ 18 years of age must sign a written informed consent. For patients < 18 years old, the patient's parents or legal guardians must sign a written informed consent, unless the patient is an emancipated minor. Childhood Assent, when age appropriate as per institutional guidelines, should be signed by the participating patient. Consent may be obtained virtually, as per institutional guidelines.

Exclusion Criteria:

* Significant organ dysfunction, not meeting inclusion criteria.
* Pediatric subjects who are considered wards of some entity
* Pregnancy or Breast-Feeding
* Pregnant or breast-feeding woman will not be entered on this study due to risks of fetal and teratogenic adverse events as seen in animal/human studies.
* Concomitant Medications:
* Growth factor: Growth factors that support platelet or white cell number of function must not have been administered within the past 7 days.
* Investigational Drugs: Patients who are currently receiving another investigational drug. (Please refer to Prior Therapy, section 2.1.5)
* Anti-cancer Agents: Patients who are currently receiving other anti-cancer agents. (Please refer to Prior Therapy, section 2.1.5.1)
* Medication Allergy:

  1. Allergy or intolerance to agents on this protocol: irinotecan, temozolomide, or eribuin
  2. Allergy to cephalosporins, without a reasonably available antibiotic alternative
* Infection: Patients who have uncontrolled infection, positive blood cultures within the past 48 hours, or receiving treatment for Clostridium difficile infection.

Ages: 1 Year to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-08-16 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion; an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Fiorela Hernandez Tejada, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org